CLINICAL TRIAL: NCT01148433
Title: Quality of Life With TESTIM® in Testosterone Replacement Therapy for Male Patients With Hypogonadism
Brief Title: Quality of Life With TESTIM®
Acronym: LIFE
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: FE999303 CS01
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TESTIM® - drug given by prescription: Male patients with Hypogonadism

SUMMARY:
The present non-interventional study is to document the testosterone levels in patients with clinical symptoms such as loss of sexual desire indicating hypogonadism (testosterone deficiency syndrome). During testosterone replacement therapy with TESTIM®, the changes in the quality of life - especially with respect to motivation, activity and fatigue - of hypogonadal patients will be documented and correlated with the testosterone levels during the course of therapy.

ELIGIBILITY:
Inclusion Criteria:

* therapeutic need according to SPC
* written informed consent

Exclusion Criteria:

* contraindications according to SPC

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private practices
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Serum Testosterone Level | 6 months
  Measured at Visit 1 (diagnosis), Visit 3 (month 3) and Visit 4 (month 6)

SECONDARY OUTCOMES:
Quality of Life - (determined by the MFI questionnaire) | 6 months
  Determined at Visit 2 (month 0), Visit 3 (month 3) and Visit 4 (month 6)
Multidimensional Fatigue Inventory (MFI) - (based on 20 questions regarding QoL) | 6 months
  Used at Visit 2 (month 0), Visit 3 (month 3) and Visit 4 (month 6)
Loss of Libido - (determined by the International Index of Erectile Function (IIEF-5) | 6 months
  Used at Visit 2 (month 0), Visit 3 (month 3) and Visit 4 (month 6)
Aging Male Scale (AMS) - (17 questions regarding the discomfort associated with testosterone deficiency) | 6 months
  Used at Visit 2 (month 0), Visit 3 (month 3) and Visit 4 (month 6)
Laboratory Parameters: PSA and Haematocrit levels | 6 months
  Measured at Visit 1 (diagnosis), Visit 3 (month 3) and Visit 4 (month 6)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (64):
- Germany (64):
  - Investigational Site, Apolda
  - Investigational Site, Aschersleben
  - Investigational Site, Bad Bergzaben
  - Investigational Site, Bad Schönborn
  - Investigational Site, Bautzen
  - Investigational Site, Helene-Weigel-Platz 10, Berlin
  - Investigational Site, Kurfürstendamm 33, Berlin
  - Investigational Site, Königin-Elisabeth-Straße 1, Berlin
  - Investigational Site, Tempelhofer Damm 227, Berlin
  - Investigational Site, Turmstraße 82, Berlin
  - Investigational Site, Wilmersdorfer Straße 62, Berlin
  - Investigational site, Bielefeld
  - Investigational Site, Bramsche
  - Investigational Site, Humboldtstraße 4, Braunschweig
  - Investigational site, Ritterbrunen 7, Braunschweig
  - Investigational Site, Dr.-Franz-Mertens-Straße 8, Bremerhaven
  - Investigational Site, Bremerhaven
  - Investigational Site, Büdingen
  - Investigational Site, Carl-von-Ossietzky-Straße 151, Chemnitz
  - Investigational Site, Clausstraße 44, Chemnitz
  - Investigational Site, Unritzstraße 21 c, Chemnitz
  - Investigational Site, Cologne
  - Investigational Site, Dortmund
  - Investigational Site, Dossenheim
  - Investigational Site, Düsseldorf
  - Investigational Site, Forchheim
  - Investigational Site, Eschersheimer Landstr. 544, Frankfurt
  - Investigational Site, Im Steinbügel 13, Frankfurt
  - Investigational Site, Freiberg
  - Investigational Site, Fulda
  - Investigational site, Gera
  - Investigational Site, Greifswald
  - Investigational Site, Halle
  - Investigational Site, Neuenfelder Straße 96, Hamburg
  - Investigational Site, Sand 35, Hamburg
  - Investigational Site, Schweriner Straße 25, Hamburg
  - Investigational Site, Tangstedter Landstraße 77, Hamburg
  - Investigational Site, Heilbronn
  - Investigational Site, Henningsdorf
  - Investigational Site, Hermsdorf
  - Investigational Site, Kamenz
  - Investigational Site, Kulmbach
  - Investigational Site, Landsberg/Lech
  - Investigational Site, Langenfeld
  - Investigational Site, Lübeck
  - Investigational Site, Mühlhausen
  - Investigational Site, München
  - Investigational Site, Neustadt
  - Investigational Site, Am Museumsturm 4, Nordhorn
  - Investigational Site, Osnabrücker Str. 1, Nordhorn
  - Investigational Site, Nuremberg
  - Investigational Site, Offenbach
  - Investigational Site, Paderborn
  - Investigational Site, Pulheim
  - Investigational Site, Ribnitz-Damgarten
  - Investigational Site, Rostock
  - Investigational Site, Rottweil
  - Investigational Site, Rüttenscheid
  - Investigational Site, Schwerte
  - Investigational Site, Tostedt
  - Investigational Site, Tönisvorst
  - Investigational Site, Weinheim
  - Investigational Site, Wilhelmshaven
  - Investigational Site, Wolfsburg